CLINICAL TRIAL: NCT05506930
Title: Intrathecal Morphine Versus Bilateral Quadratus Lumborum Blocks for Perioperative Analgesia in Pediatric Patients Undergoing Open Lower Abdominal Procedures: A Prospective Randomized Trial
Brief Title: ITM vs QL for Pediatric Open Lower Abdominal Procedures
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The study was stopped early based on the anecdotal evidence from a surgeon who felt one group was experiencing more side effects than the other. Exposing pediatric patients who would be assigned to the inferior arm was difficult to justify ethically.
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Natalie Barnett, Principal Investigator, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00121082
Record Dates: First submitted 2022-08-12; First posted 2022-08-18 (Actual); Results first posted 2025-04-15 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Pain Control; Ureteral Reimplantation; Pediatrics; Intrathecal Morphine
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant
Masking Description: The patient and their parent/guardians will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intrathecal Morphine (Active Comparator): Intrathecal Morphine: spinal (neuraxial) dose of preservative free morphine (duramorph), usually about 4-5mcg/kg
  Interventions: Drug: Intrathecal Morphine
- quadratus lumborum block (Active Comparator): Quadratus Lumborum Block: peripheral nerve block utilizing ropivacaine 0.2%, usually about ½ mL per kg per side (total dose approximately 1mL/kg).
  Interventions: Drug: Quadratus lumborum block

INTERVENTIONS:
Drug: Intrathecal Morphine — One group of subjects will receive intrathecal morphine: spinal (neuraxial) dose of preservative free morphine (Duramorph), usually about 4-5mcg/kg. This is injected into the cerebrospinal fluid under sterile technique by a pediatric anesthesiologist while the subject is already under general anesthesia. This procedure is well-described in the pediatric population and used regularly for postoperative pain relief for a variety of procedures including ureteral reimplantation.
  Other Names: ITM
  Arms: Intrathecal Morphine
Drug: Quadratus lumborum block — The second group of subjects will have bilateral quadratus lumborum blocks: peripheral nerve block utilizing ropivacaine 0.2%, usually about ½ mL per/ kg per side (total dose approximately 1mL/kg). This is injected in the subject's flank in the fascial plane between the quadratus lumborum muscle and the psoas muscle. Ultrasound guidance is used for needle and structure localization and this procedure is done by a pediatric anesthesiologist while the subject is already under general anesthesia. Quadratus lumborum blocks are regularly used in clinical practice for postoperative pain relief for a variety of abdominal procedures.
  Other Names: QL
  Arms: quadratus lumborum block

SUMMARY:
Patients between the ages of 12 months and 11 years who are undergoing an open lower abdominal procedure will be randomized to receive intrathecal morphine, or bilateral quadratus lumborum block. The investigators will compare the effect that intrathecal morphine and quadratus lumborum blocks have on the duration of pain control as demonstrated by charted pain scores and morphine equivalents in the first 48 hours. This study will also assess the side effects of each intervention such as nausea and vomiting, and itching.

ELIGIBILITY:
Inclusion Criteria:

* Ages 12 months to 11 years old
* Undergoing an open lower abdominal procedure

Exclusion Criteria:

* Allergy to morphine or amide local anesthetics
* Localized rash at site of planned regional anesthetic block
* Bleeding diathesis
* Spinal dysmorphism
* Previous spinal surgery with instrumentation of the lumbar spine
* Inability or unwillingness of parent or legal guardian to give informed consent.
* Prior enrollment and randomization in this study

Ages: 12 Months to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 14 (Actual)
Dates: Start 2022-08-17 (Actual); Primary Completion 2024-05-09 (Actual); Study Completion 2024-05-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Natalie Barnett, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intrathecal Morphine | Quadratus Lumborum Block
Started | 5 | 9
Completed | 5 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intrathecal Morphine | Quadratus Lumborum Block | Total
Number analyzed (Participants) | 5 | 9 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 5 (3.8) | 4.4 (2.8) | 4.607 (3.089)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 2 | 5 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 5 | 7 | 12
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 5 | 7 | 12
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Procedure Type [Count of Participants; unit: Participants]
  Laparoscopy | 0 | 1 | 1
  Ureteral Reimplantation | 5 | 7 | 12
  Enterocystoplasty | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Duration of Analgesia - Pain Score 0-10
Description: The primary endpoint will compare the effect that intrathecal morphine and quadratus lumborum blocks have on the duration of analgesia as demonstrated by charted pain scores in the first 24 hours. Pain scores were collected from the medical record on a scale from 0-10; the higher the score, the worse the outcome/pain. Time points in the 24 hours post op for each patient varied based on nursing care as the data was collected from the medical record.
Time Frame: Up to 24 hours post-op
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intrathecal Morphine | Quadratus Lumborum Block
Number analyzed (Participants) | 5 | 9
units on a scale | 1.0 (0.8) | 1.5 (1.4)

2. Secondary Outcome: Number of Participants With Side Effects of Each Intervention
Description: The secondary endpoint will assess the side effects of each intervention such as nausea and vomiting, and pruritis.
Time Frame: up to 48 hours post-operative
Measure: Count of Participants; unit: Participants
Arm/Group | Intrathecal Morphine | Quadratus Lumborum Block
Number analyzed (Participants) | 5 | 9
Participants
  Pruritis | 2 | 2
  Nausea and/or Vomiting | 4 | 3

3. Secondary Outcome: Severity of Side Effects With Each Intervention
Description: The secondary endpoint assesses the severity of side effects with each intervention such as nausea and/or vomiting, and pruritus in the patients who experienced a side effect. Parents of participants who experienced the side effects listed rated the severity of them using a Visual Analog Scale from 0-100mm. The higher the score, the worse the side effect.
Time Frame: 0-48 hours post-operatively
Population: Patients may have experienced one side effect or both, therefore there may be overlap in participant numbers reporting a score. Four unique participants in the intrathecal morphine group reported 6 instances of side effects, and 4 subjects in the QL group reported 5 instances of size effects.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intrathecal Morphine | Quadratus Lumborum Block
Number analyzed (Participants) | 4 | 4
units on a scale
  Pruritus: number analyzed (Participants) | 2 | 2
  Pruritus | 65.0 (21.2) | 30.0 (28.3)
  Nausea and/or Vomiting: number analyzed (Participants) | 4 | 3
  Nausea and/or Vomiting | 55.0 (17.3) | 60.0 (10.0)

4. Secondary Outcome: Patient/Family Satisfaction
Description: This endpoint will assess patient and family overall satisfaction with their child's pain control and experience of their child's post-op recovery. Satisfaction will be rated using VAS 0 (not satisfied) to 100 (completely satisfied).
Time Frame: up to 48 hours post-operative
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intrathecal Morphine | Quadratus Lumborum Block
Number analyzed (Participants) | 5 | 9
units on a scale
  Satisfaction with pain control | 89.0 (17.5) | 73.3 (29.6)
  Overall satisfaction | 88.0 (11.5) | 87.2 (17.5)

5. Secondary Outcome: Total Length of PACU Stay - Minutes
Description: This endpoint will assess how long the patient's PACU stay was in minutes. The longer the stay, the worse the outcome.
Time Frame: time to discharge after surgery, (an expected average length of hospital stay is approximately 2-4 days)
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Intrathecal Morphine | Quadratus Lumborum Block
Number analyzed (Participants) | 5 | 9
minutes | 42.8 (37.0) | 57.4 (37.0)

6. Primary Outcome: Duration of Analgesia - MME/kg in First 24 Hours
Description: The primary endpoint will compare the effect that intrathecal morphine and quadratus lumborum blocks have on the duration of analgesia as demonstrated by morphine milligram equivalents (MME)/kg in the first 24 hours. The higher the MME/kg, the worse the pain.
Time Frame: Up to 24 hours post-op
Measure: Mean (Standard Deviation); unit: MME/kg
Arm/Group | Intrathecal Morphine | Quadratus Lumborum Block
Number analyzed (Participants) | 5 | 9
MME/kg | 0.03 (0.06) | 0.08 (0.13)

7. Secondary Outcome: Total Length of Hospital Stay - Length of Stay, Days
Description: This endpoint will assess how long the patient's hospital stay was overall in days. The higher the number of days, the worse the outcome.
Time Frame: time to discharge after surgery, (an expected average length of hospital stay is approximately 2-4 days)
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Intrathecal Morphine | Quadratus Lumborum Block
Number analyzed (Participants) | 5 | 9
days | 1.4 (0.6) | 2.0 (1.6)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from 0-48 hours post-operatively through in-person assessments and chart review.
Arm/Group | Intrathecal Morphine | Quadratus Lumborum Block
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/9
Other Adverse Events (participants affected / at risk) | 4/5 | 4/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intrathecal Morphine (N=5) | Quadratus Lumborum Block (N=9)
Nausea and/or Vomiting (Gastrointestinal disorders) | 4 (4) | 3 (3) — Nausea and/or Vomiting
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) — Pruritus

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-07-13): https://cdn.clinicaltrials.gov/large-docs/30/NCT05506930/Prot_SAP_ICF_000.pdf